CLINICAL TRIAL: NCT07140289
Title: The Effect of Glucagon-like Peptide-1 Receptor Agonists (GLP-1 RA) on Gastric Emptying Before Elective Surgery
Brief Title: Effect of Glucagon-like Peptide-1 Receptor Agonists (GLP-1 RA) on Gastric Emptying
Status: Enrolling by invitation | Type: Observational
Sponsor: Wael Saasouh, MD (Other)
Collaborators: Wayne State University (Other)
Responsible Party: Sponsor-Investigator, Wael Saasouh, MD, Director of Research, Dept of Anesthesiology WSU-DMC, Wayne State University
Organization: Wayne State University (Other)
Other Study IDs: IRB 23-10-6273
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Gastric Emptying; Glucagon-Like Peptide-1 Receptor Agonists; Intermittent Fasting; Intraoperative Complication Due to Anesthesia; Respiratory Aspiration of Gastric Contents
MeSH Terms: conditions — Intermittent Fasting; Respiratory Aspiration of Gastric Contents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Study group: Adult patients who are receiving a Glucagon-like peptide-1 Receptor Agonist and scheduled for any elective surgery or procedure under anesthesia.
  Interventions: Diagnostic Test: Ultrasound of gastric contents

INTERVENTIONS:
Diagnostic Test: Ultrasound of gastric contents — An ultrasound examination of the abdomen to observe and measure gastric contents

SUMMARY:
This study aims to assess the effect of using Glucagon-like peptide-1 receptor agonists (GLP-1) receptor agonists on gastric emptying on surgical patients and whether specific guidelines need to be established for these patients. GLP-1 receptor agonists are mainly used for the treatment and mitigation of obesity and metabolic syndromes. One of their mechanisms of action is by delaying gastric emptying, hence increasing satiety. However, patients need to abstain from eating for a set amount of time before surgery to reduce the risk of aspiration. Hence patients who use GLP-1 receptor agonists may need more time to abstain eating (nil-per-os). In this study we aim to assess how much time is sufficient before surgery in these specific population of patients.

DETAILED DESCRIPTION:
Diabetes is a global health issue. It is the leading cause of death and disability worldwide. More than 1.31 billion people are projected to have diabetes in the world by 2050. Similarly in the United States total prevalence of diabetes is projected to be around 21% of the US population by 2050. Glucagon-like peptide-1 receptor agonists (GLP-1 RA), alternatively referred to as incretin mimetics, or GLP-1 analogs, constitute a category of drugs utilized for the management of type 2 diabetes mellitus and also for obesity. Glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP) are hormones known as incretin hormones. GIP hormones play a role in stimulating the release of insulin after consuming glucose, which is referred to as the incretin effect. However, in people with type 2 diabetes, this process can be diminished or absent. Pharmacological levels of GLP-1 can help restore insulin secretion in individuals with type 2 diabetes. The advantages of using this approach for treating type 2 diabetes include the slowing down of stomach emptying and the suppression of glucagon production from pancreatic alpha cells when blood sugar levels are high. Additionally, GLP-1 RAs have the potential to reduce the death of pancreatic beta cells (the cells responsible for producing insulin) while also encouraging their growth.

Recent literature have raised concerns about the potential of GLP-1 RA-induced delayed gastric emptying to heighten the risk of regurgitation and inhalation of stomach contents during instances of general anesthesia and profound sedation. The term "high-risk stomach" refers to gastric volume carrying a heightened pulmonary aspiration risk, typically defined as liquid content exceeding 1.5 ml/kg or the presence of solid matter, as commonly described in literature. Gastric ultrasound has been used as an important tool for assessing the gastric content and volume. Measurement of the antral cross-sectional area by ultrasound with subsequent calculation of gastric volume can determine the low risk or high-risk stomach accordingly (8.

In June 2023, the ASA (American Society of Anesthesiologists) released a consensus-based guideline regarding the preoperative management of patients using GLP-1 RA. The recommendation advised taking these medications either on the day before or on the day of the procedure. Patients on a weekly regimen were advised to suspend the drug for the entire week. Although there are general fasting recommendations for the general population, no fasting recommendations were provided for patients on GLP-1 RA due to insufficient supporting evidence.

This research aims to increase our understanding about the effect of use of GLP-1 RAs on gastrointestinal motility and gastric emptying. The results of this study may provide insight regarding acceptable timing of NPO (Non per oral) before surgical procedures to reduce the risk of aspiration and other related complications.

The following information will be obtained from the patients in their visit:

1. Patient's identifying information
2. Patient's age
3. Patient's gender
4. Patient's weight
5. Time of last eating or drinking
6. Consumed food in the last eating or drinking
7. Duration of fasting
8. Patient's procedure/surgery
9. Medical history, including Previous gastric resection or bypass, Previous fundoplication, Gastric band in situ, Large hiatus hernia, Pregnancy, GERD
10. Any relevant surgical history, history of substance use, and list of current medications
11. Name of GLP-1 receptor agonist drug and its brand name
12. Dose of the medication
13. Dosing interval of the medication
14. Route of administration of the medication
15. Duration of use of the medication since the first dose
16. Last time of drug administration
17. Reason for continuing GLP-1 receptor Agonist drug, including diabetes, weight loss, etc

Gastric Ultrasound Finding reporting items:

1. Whether the stomach is empty or not
2. Whether the stomach has liquid content or not
3. The right lateral antral cross-sectional area (CSA)
4. Calculated gastric volume
5. Whether the stomach has solid food

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are receiving Glucagon-like peptide-1 Receptor Agonist medication and scheduled for any elective surgery or procedure under anesthesia.
* The patient has provided informed consent for the study

Exclusion Criteria:

* Pregnant patients
* Patients with abnormal gastric anatomy like previous gastric resection or bypass( gastric band in situ, previous fundoplication, hiatus hernia
* Inability to consent
* Emergency surgery
* Cognitive impairment (due to the mixed reasons of potential misunderstanding of the aim of the study and inability to provide informed consent, potential inability to provide detailed fasting regimen before the surgery, potential for impaired use of GLP-1 agonists before the surgery)
* Terminal illness (due to the effect of chronic illness on the physiologic functions of gastrointestinal tract and gastric emptying)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgical patients undergoing procedures at the Detroit Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Gastric cross-sectional area | Preoperatively on the day of surgery (between admission to preoperative testing and start of surgical procedure).
  Ultrasound measurement of the right- lateral cross-sectional area measurement of the gastric antrum measured pre-operatively

SECONDARY OUTCOMES:
Incidence of Pulmonary Aspiration | Between induction of anesthesia and discharge (up to 4 hours) from the post-anesthesia care unit after surgery
  Documented clinical evidence of aspiration (e.g., witnessed event, presence of aspirated material in airway, or new infiltrate on chest imaging consistent with aspiration)
Incidence of Aspiration Pneumonia/Pneumonitis | Within 7 days of surgery (if data is available)
  Diagnosis based on clinical criteria (fever, leukocytosis, new infiltrate on chest X-ray, hypoxemia) and/or microbiological confirmation
Incidence of other Respiratory Complications | Within 7 days of surgery (if data is available)
  New or worsening respiratory disease (e.g., ARDS, acute respiratory failure, need for escalation of ventilatory support)
Need for Reintubation | Within 7 days of surgery (if data is available)
  Requirement for repeat endotracheal intubation due to respiratory compromise attributed to aspiration
ICU Length of Stay | Up to hospital discharge (up to 30 Days)
  Number of days in ICU following aspiration event (up to 30 days)
Hospital Length of Stay | Up to 30 days
  Number of days in hospital following aspiration event
Mortality | Within 30 days of surgery (if data is available)
  All-cause mortality within 30 days of aspiration event
Other Medical Complications | Within 7 days of surgery (if data is available)
  New onset infection (e.g., sepsis), fever, or other systemic complications following aspiration
Hypoxemia | Between emergence from anesthesia and discharge from the post-anesthesia care unit after surgery
  Oxygen saturation <90% requiring intervention (supplemental O₂, airway support)
Reintubation or Unplanned Airway Intervention | Within 7 days of surgery (if data is available)
  Requirement for repeat endotracheal intubation or advanced airway management due to respiratory compromise attributed to aspiration
Postoperative Anesthetic Respiratory Complications | Between emergence from anesthesia and discharge from the post-anesthesia care unit after surgery
  Composite of events including laryngospasm, bronchospasm, upper airway obstruction, or need for noninvasive ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Detroit Medical Center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No